CLINICAL TRIAL: NCT06826326
Title: A 'Proof of Concept' Study to Identify Neural Target Engagement of Escitalopram in Adolescents With Autism Spectrum Disorder
Brief Title: Neuroimaging of Escitalopram in Autism Spectrum Disorder
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Kathryn Unruh (Other)
Responsible Party: Sponsor-Investigator, Kathryn Unruh, principal investigator, University of Kansas
Organization: University of Kansas (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STUDY00160812
Record Dates: First submitted 2025-02-03; First posted 2025-02-13 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder
Keywords: escitalopram; autism spectrum disorder; repetitive behavior; fMRI
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Escitalopram then Placebo (Experimental): participants will receive escitalopram during visit 2 and placebo during visit 3
  Interventions: Drug: Escitalopram 10mg; Drug: Placebo
- Placebo then Escitalopram (Experimental): participant will receive placebo during visit 2 and escitalopram during visit 3
  Interventions: Drug: Escitalopram 10mg; Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram 10mg — oral administration of escitalopram 10 mg
Drug: Placebo — Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the acute effects of escitalopram (Lexapro®) on select brain networks during task-based functional magnetic resonance imaging (fMRI) in adolescent individuals with autism spectrum disorder (ASD). We hope to learn more about the acute effects of escitalopram and how it might be used to treat inflexible thinking or rigid-compulsive behavior that can be associated with restricted and repetitive behaviors in adolescents with ASD.

Participants will:

* Attend 3 visits to complete tests of thinking abilities and fill out surveys about their health and behavior
* Be randomly assigned to receive escitalopram at one of the first two visits after screening and a placebo at the other visit.
* Complete a reward-based task that tracks eye movement, either during MRI or in laboratory environment.

DETAILED DESCRIPTION:
This study is a randomized placebo-controlled, cross-over design evaluating the effects of escitalopram (Lexapro®) on behavioral inflexibility in autism spectrum disorder (ASD). The trial will be conducted on individuals with ASD aged 12-17 years old.

The neural target engagement experiment will use a randomized, placebo-controlled, cross-over design. Within one month after completing the Screening Visit, participants will be randomized by the statistician, in communication with the site pharmacy, to take a single dose of either escitalopram 10 mg or placebo (Visit 2) three hours before beginning the functional MRI. A minimum of one week later (Visit 3), participants will take the other medication (placebo or escitalopram 10 mg) three hours before beginning the functional MRI.

The primary objective of this 'proof of concept' study is to identify neural target engagement of escitalopram in adolescents with ASD.

Primary Objective 1. Neural target engagement: Evaluate the impact of a single dose of escitalopram 10 mg versus placebo, in a cross-over design, on blood-oxygen-level dependent (BOLD) activation during a rewarded inhibitory control functional MRI (fMRI) task that has previously shown to be sensitive to individual differences in restricted and repetitive behavior (RRB) severity in ASD (preliminary data).

Primary Objective 2. Behavioral target engagement-inhibitory control: Evaluate the impact of a single dose of escitalopram 10 mg versus placebo, in a cross-over design, on behavioral inflexibility during a rewarded inhibitory control task that has previously shown to be sensitive to individual differences in RRB severity in ASD (preliminary data).

Secondary Objective 1. Neural target engagement: Evaluate the impact of a single dose of escitalopram 10 mg versus placebo, in a cross-over design, on blood-oxygen-level dependent (BOLD) activation during a rewarded prosaccade functional MRI (fMRI) task.

Secondary Objective 2. Behavioral target engagement-prosaccades: Evaluate the impact of a single dose of escitalopram 10 mg versus placebo, in a cross-over design, on reflexive motor behavior during a rewarded prosaccade task.

ELIGIBILITY:
Inclusion Criteria:

All participants must meet all inclusion criteria:

1. Participant must be at least 12 years old and no greater than 17 years old.
2. A parent or guardian must sign an informed consent document indicating understanding the protocol and procedures and willingness to participate in full. Signed assent indicating understanding and willingness to participate is required of participants under 18 years of age (all participants).
3. Participant must have a diagnosis of Autism Spectrum Disorder, according to DSM-5 criteria, made by a licensed study psychiatrist or psychologist and supported by the Autism Diagnostic Observation Schedule 2 (ADOS-2) completed at screening or within the past 12 months by an appropriately trained professional.
4. Participant must have a non-verbal IQ of greater than or equal to 70 as determined by the 4-subtest Wechsler Abbreviated Scale of Intelligence.
5. Participant must be able to speak and understand English in order to complete study measures.
6. Participant must live with a parent, primary caregiver, or other adult informant who can complete study measures on the basis of spending an average of at least 4 hours per day with the participant.
7. Parent, primary caregiver, or other adult informant must speak and understand English to complete study measures.
8. Participant must be able to self-administer study medication or have parent/caregiver be able to administer study medication.
9. Participant must be able to swallow study medication whole with liquid.
10. Participant or legally acceptable representative must be willing to continue current medication(s) and behavioral intervention(s) and to not add or change medication(s) or behavioral intervention(s) over the full course of the study.

Exclusion Criteria

Any potential subject who meets any of the following criteria will be excluded from participating in the study unless otherwise specified:

1. Participant is judged by the Investigator to be unable to perform or comply with all study specific requirements.
2. Participant is an employee of an investigator with direct involvement in the proposed study or other studies under the direction of a study investigator, or is a family member of an investigator.
3. Participant has a history of any severe or unstable psychiatric condition (e.g., schizophrenia or other psychotic disorder, bipolar disorder, major depressive disorder) that, in the opinion of the Investigator, could confound the interpretation of the study results or put the subject at undue risk. An acute episode of a mood disorder will be considered exclusionary; a participant with a history of mild to moderate mood disorder may be included in the study under the discretion of the Investigator. Other stable psychiatric conditions are permitted at the discretion of the Investigator (e.g., attention deficit hyperactivity disorder, generalized anxiety disorder, etc.).
4. Subject has a current or recent history of clinically significant suicidal ideation within the past 6 months, corresponding to a score of 3 or higher (active suicidal ideation with some intent to act, without specific plan) on the Columbia Suicide Severity Rating Scale (C-SSRS), or a history of suicidal behavior within the past year, as validated by the C-SSRS at any study visit. In the case that a screened participant exhibits concerns on the C-SSRS that would preclude study participation, the study safety plan outlined in 1.3 Potential Risks will be followed.
5. Subject has met DSM-5 criteria for a substance abuse disorder within the last 6 months prior to Screening, except for disorders related to caffeine or nicotine.
6. Subject is taking an MAO inhibitor, serotonergic reuptake inhibitor, or serotonergic-norepinephrine reuptake inhibitor or has taken any of these medications within the past 90 days.
7. Subject is taking a psychotropic medication or has taken this medication within the past 90 days.
8. Subject has received electroconvulsive therapy (ECT) in the last 6 months.
9. Subject has received new-onset psychotherapy or has had a change in the intensity of psychotherapy within the 2 months prior to Screening.
10. Subject has known allergies, hypersensitivity, or intolerance to escitalopram or its excipients.
11. Subject has received an investigational drug or used an investigational medical device within 3 months before the planned start of study or is currently enrolled in an investigational study.
12. Subject has a body mass index (BMI) <17 at Screening.
13. Subject has a known history of long QT syndrome or family history of sudden death.
14. Subject has a history of myocardial infarction, unstable angina, acute coronary syndrome, or cerebrovascular accident (CVA) within the last 4 months. Has greater than NYHA Class 2 congestive heart failure or Class 2 angina pectoris, sustained ventricular tachycardia (VT), ventricular fibrillation, torsade de pointes, or syncope due to an arrhythmia.
15. Subject has a history of neuroleptic malignant syndrome/serotonin syndrome.
16. Subject has had a seizure within the past 12 months. Individuals with seizure disorders who are on stable seizure medications (i.e., without seizures in past 12 months) are permitted at the discretion of the Investigator.
17. Subject is pregnant or breast-feeding, or planning to become pregnant or breastfeed while enrolled in this study or within 3 months after the last dose of study drug.
18. Subject has current evidence, or a history within the previous 3 months prior to screening, of a serious and/or unstable neurologic, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical disorder, that, in the opinion of the Investigator, would jeopardize the safe participation of the subject in the study.
19. Subject has a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the Investigator, is considered cured with minimal risk of recurrence).
20. Subject has a known history of a positive hepatitis C virus (HCV) or human immunodeficiency virus (HIV) test.
21. Subject has COVID-19 vaccination status that prevents them from participating at study locations according to the institutional, local, or state guidelines at that study site.
22. Subject has other clinically significant laboratory abnormalities that, in the opinion of the Investigator, would jeopardize the safe participation of the study subject.
23. Subject is free of any medication that may affect cognitive or motor performance, as evaluated by the Investigator.
24. Subject or immediate family member has a history of kidney disease.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Rewarded Antisaccade task | At Visit 2 (1 day to 1 month after Screening/Visit 1) and Visit 3 (5 days to 3 weeks after Visit 2)
  During the rewarded antisaccade task (R-ANTI), participants are instructed to look away from a peripheral target and to the mirror location in the opposite hemifield (antisaccade) and avoid looking toward the peripheral target (prosaccade). Two trial types are presented: reward and no-reward. Number of prosaccades is compared between reward and no-reward trial types.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn E Unruh, PhD, Principal Investigator — University of Kansas
Locations (1):
- Hoglund Biomedical Imaging Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No